CLINICAL TRIAL: NCT07051512
Title: Effect of Different Doses Of Intrathecal Dexmedetomidine In Combination With Bupivacaine On Spinal Anesthesia And Its Postoperative Analgesic Effects In Patients Undergoing Infra-Umbilical Surgeries.
Brief Title: Effect of Different Doses Of Intrathecal Dexmedetomidine In Combination With Bupivacaine On Spinal Anesthesia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Marwa Gamal Abd-Elnaby Elakraa, Resident, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 36264MS266/7/23
Record Dates: First submitted 2025-06-26; First posted 2025-07-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-06

CONDITIONS: Spinal Anesthesia Evaluation; Analgesic; Intrathecal Anesthesia
Keywords: Dexmedetomidine; Bupivacaine; Spinal Anesthesia; Postoperative Analgesic; Infra-Umbilical Surgeries
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: All techniques will be performed by one anesthesiologist while the measurements will be taken by another anesthesiologist who is blinded to the study groups and has no subsequent involvement in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group (I):dexmedetomidine 4μg (Experimental): Group (I): in this group patients will receive (0.5% hyperbaric bupivacaine 12.5 mg + dexmedetomidine 4μg)
  Interventions: Drug: dexmedetomidine 4μg
- Group (II): dexmedetomidine 8 μg (Experimental): Group (II): in this group patients will receive (0.5% hyperbaric bupivacaine 12.5 mg + dexmedetomidine 8 μg)
  Interventions: Drug: dexmedetomidine 8 μg
- Group (III): dexmedetomidine 10 μg (Experimental): Group (III): in this group patients will receive (0.5% hyperbaric bupivacaine 12.5 mg + dexmedetomidine 10 μg
  Interventions: Drug: dexmedetomidine 10 μg

INTERVENTIONS:
Drug: dexmedetomidine 4μg — patients received (0.5% hyperbaric bupivacaine 12.5 mg + dexmedetomidine 4μg)
  Arms: Group (I):dexmedetomidine 4μg
Drug: dexmedetomidine 8 μg — patients received (0.5% hyperbaric bupivacaine 12.5 mg + dexmedetomidine 8 μg)
  Arms: Group (II): dexmedetomidine 8 μg
Drug: dexmedetomidine 10 μg — patients received (0.5% hyperbaric bupivacaine 12.5 mg + dexmedetomidine 10 μg).
  Arms: Group (III): dexmedetomidine 10 μg

SUMMARY:
This study is designed to assess the efficacy of different doses of dexmedetomidine in combination with intrathecal hyperbaric bupivacaine on spinal anesthesia and its postoperative analgesic characteristics on patients undergoing infra-umbilical procedures.

Primary outcome:

To ascertain a safe intrathecal dexmedetomidine dose for patients undergoing elective lower abdominal and lower limb surgeries

Secondary outcomes:

Assessment of level of sedation. Assessment of hemodynamic parameters (Blood Pressure -Heart Rate). Assessment of level of sensory & motor block. Assessment of pain.

DETAILED DESCRIPTION:
Pain is an unpleasant sensory and emotional experience associated with actual or potential tissue damage. A pain free and stress free postoperative period helps in early mobilization and recovery of surgical patients, thereby reducing morbidity. Intraoperative and postoperative pain relief is a fundamental component of anesthesia. Accordingly, anesthesiologists constantly strive to offer the best possible anesthetic technique with emphasis on minimum adverse effects and satisfactory perioperative analgesia. Spinal anesthesia is a preferred technique to administer anesthesia for infraumbilical operations. However, postoperative pain control is a matter of concern with spinal anesthesia using only local anesthetics, as the analgesic effect lasts for a relatively short duration. Thus, early analgesic intervention is needed in the postoperative period.

Various adjuvants, such as opioids, epinephrine, neostigmine, magnesium, midazolam, ketamine, clonidine, have been used with intrathecal local anesthetics in attempts to prolong analgesia and reduce the incidence of adverse events. In recent years, α2-adrenergic receptor agonists have gained popularity as an important adjunct in anesthetic practice, whether it be general or regional anesthesia.

Dexmedetomidine is selective alpha-2 agonist with favorable analgesic, sedative, anxiolytic, and sympatholytic features. Researchers have used dexmedetomidine intrathecally in varying doses with varying results. Despite extensive research, no consensus on optimal dose of intrathecal dexmedetomidine exists, since with higher doses there is better intraoperative and post-operative analgesia, but there is an increased likelihood of hemodynamic disturbances.

This prompted us to conduct this research to study varying doses of intrathecal dexmedetomidine to compare the prolongation of sensory and motor block duration with dosage ranging from as low as 4 μg to as high as 10 μg as adjuvant along with 0.5% hyperbaric bupivacaine. Anticipated benefits/outcomes included prolongation of sensory and motor block with reduced/ delayed need of rescue analgesics in the post-operative period and with reduced intraoperative and post-operative side effects.

This study is designed to assess the efficacy of different doses of dexmedetomidine in combination with intrathecal hyperbaric bupivacaine on spinal anesthesia and its postoperative analgesic characteristics on patients undergoing infra-umbilical procedures.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years of either sex.
* American Society of Anesthesiologists physical status I and II.
* undergoing elective lower abdominal and lower limb surgeries under planned subarachnoid block.

Exclusion Criteria:

* patient refusal
* contraindication to subarachnoid block (hypersensitivity to the drugs - infection at the site of injection)
* significant comorbid conditions like congestive heart failure, coagulopathy, heart block
* pregnancy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
intrathecal dexmedetomidine dose | 2 hours
  To ascertain a safe intrathecal dexmedetomidine dose for patients undergoing elective lower abdominal and lower limb surgeries.3. The sensory block level will be assessed at 5 min , 20 min after administration of spinal anesthesia and every 15 min postoperative until two segment sensory regression.
A safe intrathecal dexmedetomidine dose for patients | Intraoperative during 2 hours
  To ascertain a safe intrathecal dexmedetomidine dose for patients undergoing elective lower abdominal and lower limb surgeries

SECONDARY OUTCOMES:
pain by Visual analogue scale | 24 hours postoperatively.
  The pain onset time in the postoperative period will be assessed using Visual analogue scale hourly for the first 4hours, then every 4 hours for the next 8 hours, and at 24 hours postoperatively.
intraoperative sedation level using the Ramsay sedation scale | 24 hours post-spinal injection
  The intraoperative sedation level of the patients will be assessed using the Ramsay sedation scale. The patient will be considered to be sedated if the Ramsay sedation scale score was ≥2 and will be assessed hourly till 4 hours after surgery and then at 8 hours, 12 hours and 24 hours post-spinal injection.

CONTACTS AND LOCATIONS:
Overall Officials: Marwa Elakraa, Resident, Principal Investigator — Tanta University
Locations (1):
- Tanta University, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided